CLINICAL TRIAL: NCT03771872
Title: Effects of Virtual Prism Adaptation Therapy in Stroke Patients With Hemispatial Neglect
Brief Title: Virtual Prism Adaptation Therapy on Hemispatial Neglect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment of subjects has been difficult.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bundang Rusk Rehabilitation Specialty Hospital (Unknown)
Responsible Party: Principal Investigator, Won-Seok Kim, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-0154-004
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Recovery of Function; Rehabilitation; Perceptual Disorders; Virtual Reality Exposure Therapy
MeSH Terms: conditions — Stroke; Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Prism Adaptation Therapy (Experimental): This group will be provided with real virtual prism adaptation therapy. In the real therapy session, the hand trajectory will deviate to the right side in the virtual reality. The deviation angle will be adjusted according to the subject's adaptation. 20min-session will be provided twice a day for 5 days, then the total 10 sessions of therapy will be provided.
  Interventions: Device: Virtual Prism Adaptation Therapy
- Sham Therapy (Sham Comparator): The therapy is the same as the real virtual prism adaptation therapy, but there will be no deviation of the hand trajectory in the virtual reality.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Virtual Prism Adaptation Therapy — Hand trajectory will deviate to the right side in the virtual reality.
  Arms: Virtual Prism Adaptation Therapy
Device: Sham Therapy — The therapy is the same as the real virtual prism adaptation therapy, but there will be no deviation of the hand trajectory in the virtual reality.
  Arms: Sham Therapy

SUMMARY:
The purpose of this study is to investigate the effect of virtual prism adaptation therapy on hemispatial neglect in chronic stroke patients. This study is the randomized, double-blind, sham-controlled, cross-over design. Total 10 patients will be allocated randomly to either real virtual prism adaptation therapy or sham therapy with the wash-out period of more than 2 weeks. Two sessions (20min/session) per day, for 5days (total 10 sessions) will be provided. Behavioral outcomes will be measured before and after completing a total of 10 sessions therapy.

ELIGIBILITY:
Inclusion Criteria:

* 3 months after stroke onset
* 2 or more tests indicative of hemispatial neglect in following 3 tests: 1)line bisection test, 2)Albert's test, 3)Drawing test.
* Ability to recognize the target object, hand trajectory in the immersive virtual reality
* 16 points or more in the Korean version of mini-mental state examination

Exclusion Criteria:

* Previous stroke or traumatic brain injury history
* Can not cooperate during the therapy, due to delirium or aphasia
* Unstable medical conditions
* Severe psychiatric symptoms that interfere with the therapy participation (e.g. severe depression, agitation, psychotic symptoms)
* Pregnancy
* Can not maintain sitting posture

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Behavioral Inattention Test (BIT) Score | Change from Baseline at 5 days
  Range: 0(best) to 227(worst)

SECONDARY OUTCOMES:
BIT Conventional subtest score (BITC) | Change from Baseline at 5 days
  Range: 0(best) to 146(worst)
BIT Behavioral subtest score (BITB) | Change from Baseline at 5 days
  Range: 0(best) to 81(worst)
Comb and Razor Test | Change from Baseline at 5 days
  Range: 0% deviation (best) to 100% deviation (worst)
Catherine Bergego Scale (CBS) | Change from baseline at 5 days
  Range: 0 (best) to 30 (worst)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Bundang Rusk Rehabilitation Specialty Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do